CLINICAL TRIAL: NCT01881061
Title: Lung Sonography in Patients With Acute Respiratory Distress Syndrome in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Serafim Nanas, Professor of Critical Care Medicine, University of Athens
Other Study IDs: UOA-US-2010
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: ARDS
Keywords: Sonography; ICU; PEEP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the role of lung sonography during different PEEP settings in ICU patients with ARDS.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a clinical syndrome that often occurs in critically ill patients.

Patients with ARDS invariably require mechanical ventilation to improve oxygen transport. An improvement in oxygenation can be obtained by an increase in positive end-expiratory pressure (PEEP).

In critically ill patients with ARDS, lung imaging is been held by the use of chest radiography and the "gold standard" technique, Computed Tomography (CT).

We designed an observational study in which we included patients under mechanical ventilation admitted in our ICU. In all patients PEEP changes were applied and lung sonography was performed.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with ARDS admitted in ICU of Evangelismos Hospital
* length of stay > 48 hours

Exclusion Criteria:

* age < 18 years
* emphysema fractures or skin lesions that do not allow the implementation of lung sonography
* BMI > 35 kg/m2
* length of stay < 48 hours

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU population
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Non aerated lung area changes | 20 min after PEEP trial

SECONDARY OUTCOMES:
Arterial oxygen and carbon dioxide partial pressure | 20 min after PEEP trial

CONTACTS AND LOCATIONS:
Overall Officials: Serafim Nanas, MD, Study Chair — University of Athens
Locations (1):
- First Critical Care Unit, Evaggelismos Hospital, School of Medicine, University of Athens, Athens, Attica, Greece

REFERENCES:
- [Result] Stefanidis K, Dimopoulos S, Tripodaki ES, Vitzilaios K, Politis P, Piperopoulos P, Nanas S. Lung sonography and recruitment in patients with early acute respiratory distress syndrome: a pilot study. Crit Care. 2011 Aug 4;15(4):R185. doi: 10.1186/cc10338. PMID 21816054